CLINICAL TRIAL: NCT01153906
Title: Post-marketing Safety Study of Autoimmune Diseases Following Cervarix® Vaccination in Females Aged 9-25 Years in the US
Brief Title: Post-marketing Safety Study of Autoimmune Diseases Following Cervarix® Vaccination
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113522
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-09

CONDITIONS: Infections, Papillomavirus
Keywords: autoimmune diseases; HPV vaccine; papillomavirus; human papillomavirus; HPV
MeSH Terms: conditions — Papillomavirus Infections; Autoimmune Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Exposed cohort: Females 9-25 years of age, who received at least one dose of Cervarix® as part of their routine health care.
  Interventions: Other: Data collection
- Unexposed cohort: Females 9-25 years of age, who did not receive Cervarix®
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — New onset of cases for endpoints of interest in the targeted population will be identified from ambulatory and inpatient electronic administrative data and will be confirmed by blinded review of the medical record by an Endpoint Adjudication Committee (EAC) that will confirm the AID case and will assess whether the onset of disease falls within the observation period. Fibromyalgia and psoriasis, for which a high number of cases are expected, will be identified from the electronic administrative data only.

SUMMARY:
The purpose of this post-marketing study is to evaluate the incidence of autoimmune diseases (AIDs) following females who have received at the least the first dose of Cervarix® as part of their routine health care.

ELIGIBILITY:
Inclusion Criteria:

Both cohorts:

* Have complete medical insurance coverage and pharmacy benefits.
* Enrolled female health plan members for at least one year prior to study entry.
* Age between 9 and 25 years at study entry.

Exposed cohort:

• Subjects who have received at least one dose of Cervarix®, with or without any other US age-appropriate recommended vaccines.

Unexposed cohort:

• No further specific inclusion criteria

Exclusion Criteria:

Both cohorts:

• Subjects with a diagnostic code of any of the AID endpoints of interest during the one year prior to the index date.

Exposed cohort:

• Subjects who received any dose of Gardasil® prior to the first dose of Cervarix®.

Unexposed cohort:

• Subjects who receive any dose of Cervarix® prior to the index date.

Ages: 9 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females between the ages of 9-25 years
Sampling Method: Probability Sample
Enrollment: 1516 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of new cases of confirmed neuroinflammatory autoimmune diseases and other autoimmune diseases. | During the 12-month period following administration of at least the first dose of Cervarix® among the exposed cohort and during an equivalent time period among the unexposed cohort.

SECONDARY OUTCOMES:
Occurrence of new cases of confirmed systemic autoimmune diseases, organ-specific T-cell mediated autoimmune disease and organ-specific antibody-mediated autoimmune diseases. | During the 12-month period following administration of at least the first dose of Cervarix® among the exposed cohort and during an equivalent time period among the unexposed cohort.
Occurrence of new cases of fibromyalgia | During the 12-month period following administration of at least the first dose of Cervarix® among the exposed cohort and during an equivalent time period among the unexposed cohort.
Occurrence of new cases of psoriasis | During the 12-month period following administration of at least the first dose of Cervarix® among the exposed cohort and during an equivalent time period among the unexposed cohort.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilmington, Delaware, United States